CLINICAL TRIAL: NCT04007822
Title: Evaluation of the 'Pain Navigator Tool' During Physiotherapy Consultations in Patients With Chronic Low-back Pain: a Service Evaluation Trial.
Brief Title: Pain Navigator Tool for Self-management in Back Pain: PATiENCe Trial
Acronym: PATiENCe
Status: Withdrawn | Type: Observational
Why Stopped: Unable to collect data due to COVID19
Sponsor: Glasgow Caledonian University (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Other Study IDs: 260667
Record Dates: First submitted 2019-05-23; First posted 2019-07-05 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Chronic Low-back Pain; Self Efficacy; Therapeutic Alliance; Communication
Keywords: low back pain; self-efficacy; therapeutic alliance; communication
MeSH Terms: conditions — Communication; Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physiotherapists: Physiotherapists will be recruited using the following inclusion criteria: (1) two years of experience in treating patients with chronic pain, (2) currently working in an MSK outpatient clinic and (3) able to read and speak English to a level allowing satisfactory completion of the study procedures. There are no exclusion criterium. Potential participants will be recruited through the relevant gatekeeper. The gatekeeper will be responsible of forwarding the participant information sheet and consent form to the physiotherapists. Physiotherapists will be asked to demonstrate their interest by replying to the email. Any questions will be answered by the research team via email or phone.
  Interventions: Behavioral: Pain Navigator Tool

INTERVENTIONS:
Behavioral: Pain Navigator Tool — The Pain Navigator Tool (PNT) was developed recently with the aim to empower patients through helping them to discuss their main concerns about pain, and to help therapists to prioritise addressing these concerns (Blomkvist et al., 2018). The initial pilot study with this tool improved the content of the consultations and patient engagement, and led to better patient-therapist interaction in a small population of healthcare providers and patients (Blomkvist et al., 2018). As it endeavours to facilitate the implementation of self-management in patients with chronic pain, the PNT aligns with the Scottish Intercollegiate Guidelines Network (SIGN) guideline for chronic pain and the Scottish Government's strategic vision (Scottish Government, 2011; SIGN, 2013).

SUMMARY:
This study explores the experience of physiotherapists and patients using the Pain Navigator Tool during outpatient musculoskeletal consultations.

DETAILED DESCRIPTION:
Chronic pain is the largest cause of disability globally and affects up to 28 million people in the UK alone. Nearly half of those who experienced chronic pain in Europe reported receiving insufficient pain management. Conventional treatments commonly used in physiotherapy continue to show only moderate effects in pain management. A potential avenue to improve the global effect of treatments may lie in exploring non-specific treatment moderators such as the therapeutic alliance (TA). Findings suggest that it is linked with engagement in rehabilitation and is a strong predictor of treatment outcomes and adherence. This study aims to evaluate and compare the quality of practice with or without the Pain Navigator Tool (PNT). Understanding the impact of the PNT on therapeutic alliance would open an avenue to improve chronic pain management, reduce healthcare-related expenses and increase the quality of life in the population studied. In addition, exploring the experience of the physiotherapists with using the PNT will provide an in-depth understanding of its use and applicability in similar settings.

The aims of this study are to:

1. To evaluate and compare the quality of practice with or without the PNT in patients with chronic low-back.
2. To collect preliminary data on the usability and practicality of the PNT for physiotherapists.

ELIGIBILITY:
Inclusion Criteria:

Patient:

* Participant aged >18 years
* Low-back pain for more than three months
* Able to read and speak English to a level allowing satisfactory completion of the study procedures
* Initial appointment with a participating physiotherapist

Physiotherapist:

* 2 years of experience in treating patients with chronic pain
* Currently working in an MSK outpatient clinic
* Able to read and speak English to a level allowing satisfactory completion of the study procedures

Exclusion Criteria:

Patient:

* Low-back pain is not the primary reason for physiotherapy appointment
* Return appointment with physiotherapist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physiotherapists working in an MSK outpatient clinic and are able to read and speak English to a level allowing satisfactory completion of the study procedures.
  Patients with chronic low back pain attending an MSK outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Semi-Structured Interview | 4 weeks
  Semi-structured interviews with the participating physiotherapists will explore the experience using the PNT.
Change in the Health Care Providers Pain and Impairment Relationship Scale | 0 weeks, 4 weeks and at 1 month follow-up
  The HC-PAIRS is selected to assess the pain-related attitudes and beliefs of physiotherapists. It is a validated tool with adequate psychometric properties and has already been used in the selected population. It measures attitudes and beliefs on a scale of 13 to 91 with higher scores on this scale indicating stronger beliefs that LBP validates disability.
The Pain Self-Efficacy Questionnaire | 4 weeks
  The PSEQ is selected to capture the patients' levels of confidence in carrying out day-to-day tasks despite the presence of pain. It assesses the confidence of people with any type of chronic pain in activity despite pain. It covers enjoying activities, household daily activities, social life, coping in general, work, leisure activities, coping with pain without medication, accomplishing goals, living a normal lifestyle, and becoming more active, all 'despite pain'. Each is rated on a 7 point scale from 0 = not at all confident to 6 = completely confident. The total score, ranging from 0 to 60, is calculated by adding the scores for each item. Higher scores reflect stronger self-efficacy beliefs.

SECONDARY OUTCOMES:
Change in the Pain Understanding and Confidence Questionnaire | 0 weeks, 4 weeks and at 1 month follow-up
  The PUnCQ is a two-part questionnaire assessing students' knowledge and understanding of pain alongside their confidence in applying this understanding. The questionnaire consists of a chronic pain case vignette, with the first set of questions consisting of a 12-item multiple choice questionnaire, assessing knowledge and understanding in the context of the vignette. The second part of the tool is a 21-item Likert scale ranging from "not at all confident" (0) to "no problem!" (10), with a higher score indicating a higher self-perceived confidence in applying this understanding. Correct answers in the Understanding section were awarded a score of 1, and incorrect a score of 0, with a total accumulated to give a score for each participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Glasgow Caledonian university, Glasgow, Strathcylde, United Kingdom

IPD SHARING:
Plan to Share IPD: No